CLINICAL TRIAL: NCT05734352
Title: Patient Experiences of the CVA Care Program on the Stroke Unit
Brief Title: Patient Experiences on the Stroke Unit
Acronym: BIC4CVAPREMS
Status: Enrolling by invitation | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Other Study IDs: BIC4STROKEPREMS
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Completion of questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Completion of the patient reported experience measurements (PREMs) questionnaire

SUMMARY:
In this study we want to develop and validate a PREM for patient with ischemic stroke.

DETAILED DESCRIPTION:
Patient Reported Experience Measures (PREMs) assess patient's perception of health care. Currently, there is no suitable PREM tool for patients with ischemic stroke. Therefore, we aim to develop and validate a PREM for this patient population. This PREM will be validated in a multicentre study, in 10 Flemish hospitals. We want to investigate the feasibility of our new questionnaire, as well as the usefulness. In addition we well analyse the results of the questionnaires and use this information to improve the quality of the care program for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* ischemic stroke
* stayed at least one day at the stroke unit

Exclusion Criteria:

* not able to read the questionnaire
* not able to answer question orally
* are not proficient in the dutch language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Validation of a new Patient Reported Experience Measurements (PREMs) for stroke patients | 6-months
  Validation of a questionnaire which was developed based on literature and consensus meeting

SECONDARY OUTCOMES:
Patient experiences | 6-months
  How do patients experience their received care when they are admitted to the stroke unit/neurology department

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No